CLINICAL TRIAL: NCT00246402
Title: Anti-Lipolytic Strategy for HIV Lipodystrophy
Brief Title: Acipimox to Improve Hyperlipidemia and Insulin Sensitivity Associated With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Colleen Hadigan, MD MPH, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 337; R21HL073675 (NIH)
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2007-12

CONDITIONS: Insulin Resistance; Cardiovascular Diseases; Heart Diseases; HIV Infections; Hypertriglyceridemia; Hyperlipidemia
MeSH Terms: conditions — Insulin Resistance; Cardiovascular Diseases; Heart Diseases; HIV Infections; Hypertriglyceridemia; Hyperlipidemias | interventions — acipimox

INTERVENTIONS:
Drug: Acipimox

SUMMARY:
The purpose of this study is to test whether chronic administration of the drug acipimox will improve hyperlipidemia and insulin sensitivity among HIV infected patients experiencing highly active antiretroviral therapy (HAART) associated metabolic disturbances.

DETAILED DESCRIPTION:
BACKGROUND:

HIV infected patients treated with HAART are at increased risk for developing significant dyslipidemia, insulin resistance, and abnormal patterns of fat distribution. While the exact mechanism responsible for these changes is not known, there is increasing evidence that patients with HIV infection and fat redistribution have increased basal rates of lipolysis and elevated circulating free fatty acids (FFA). Patients with HIV associated lipodystrophy have increased FFA levels that correlated directly with impaired glucose metabolism and triglyceride concentrations. Furthermore, acute inhibition of lipolysis in patients with HIV lipodystrophy and insulin resistance results in improvement in insulin sensitivity. However, long-term administration of lipolytic blocking agents has not been evaluated in this patient population. Acipimox, a nicotinic acid analogue and a potent inhibitor of lipolysis, is an established therapy for dyslipidemia. In addition, through effects on lowering circulating FFA, acute administration of acipimox has been shown to improve insulin sensitivity in other populations, including lean and obese individuals and patients with type II diabetes. This study will test the hypothesis that chronic administration of acipimox will improve hyperlipidemia and insulin sensitivity among HIV infected patients experiencing HAART associated metabolic disturbances.

DESIGN NARRATIVE:

The study will be a 3-month double-blind placebo-controlled trial of 250 mg of acipimox three times daily in 30 patients with HAART lipodystrophy. The primary clinical endpoint of this study will be the change in fasting triglyceride concentration, comparing baseline values to those obtained after 3 months of acipimox or placebo. Insulin sensitivity, an important secondary endpoint, will be determined by hyperinsulinemic euglycemic clamp studies. Rates of lipolysis in the fasting state will be quantified by a 3-hour infusion of stable isotope-labeled glycerol. Indirect calorimetry will be used to assess changes in resting energy expenditure. Cross-sectional computed tomography (CT) imaging of the thigh and abdomen will allow for measurement of visceral and subcutaneous fat areas. Dual energy x-ray absorptiometry (DEXA) will be used to determine whole body fat mass.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Stable antiretroviral regimen for greater than 3 months
* Hypertriglyceridemia (fasting triglycerides greater than 150mg/dl)
* Evidence of fat redistribution (e.g., increased abdominal or cervical fat, and/or decreased subcutaneous fat of the face, arms, or legs) on physical exam

Exclusion Criteria:

* Current therapy with a lipid lowering medication (e.g., fibrates, HMG CoA reductase inhibitors, resins) or treatment with these agents in the 3 months prior to study entry
* Current use of hormone replacement therapy, oral contraceptives for women, or supraphysiologic testosterone therapy in men
* Fasting triglycerides greater than 1000mg/dl
* Active alcohol or substance abuse
* Active peptic ulcer disease
* History of renal failure or serum creatinine greater than 2.0
* Serious opportunistic infection within the 3 months prior to study entry
* Hemoglobin less than 11.0 mg/dl
* Elevated transaminase levels (AST or ALT greater than 2.5x the upper limit of normal)
* Previously diagnosed diabetes mellitus or patients receiving current treatment for diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-09; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Fasting Triglyceride Concentration (Initial, after 3 months)

SECONDARY OUTCOMES:
Insulin Sensitivity (Initial, after 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M. Hadigan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Hadigan C, Liebau J, Torriani M, Andersen R, Grinspoon S. Improved triglycerides and insulin sensitivity with 3 months of acipimox in human immunodeficiency virus-infected patients with hypertriglyceridemia. J Clin Endocrinol Metab. 2006 Nov;91(11):4438-44. doi: 10.1210/jc.2006-1174. Epub 2006 Aug 29. PMID 16940448